CLINICAL TRIAL: NCT04344184
Title: SAFEty Study of Early Infusion of Vitamin C for Treatment of Novel Coronavirus Acute Lung Injury (SAFE EVICT CORONA-ALI)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HM20018977
Record Dates: First submitted 2020-04-09; First posted 2020-04-14 (Actual); Results first posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: COVID-19; Lung Injury, Acute; Kidney Injury
MeSH Terms: conditions — COVID-19; Acute Lung Injury | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Infusion (Active Comparator): L-Ascorbic Acid (Vitamin C), intravenous infusion
  Interventions: Drug: L-ascorbic acid
- Placebo (Placebo Comparator): Dextrose 5% Water
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: L-ascorbic acid — 50 mg/kg intravenous vitamin C infusion every 6 hours for up to 96 hours
  Other Names: Vitamin C, Intravenous
  Arms: Infusion
Other: Placebo — Dextrose 5% Water
  Arms: Placebo

SUMMARY:
This study will evaluate the safety of a 96-hour intravenous vitamin C infusion protocol (50 mg/kg every 6 hours) in patients with hypoxemia and suspected COVID-19.

DETAILED DESCRIPTION:
The intravenous vitamin C treatment protocol will be comprised of four intravenous infusions a day, that is 50 mg/kg every 6 hours in patients with laboratory-confirmed SARS-CoV-2 infection manifesting COVID-19 (Novel Coronavirus Disease 2019) with hypoxemia. Treatment protocol will continue for 4 days (96 hours), and, if needed, the last study-specific bloodwork with being collected on day 7. All subjects will be followed to day 28 (phase I) and day 90 (phase II) for collection of clinical outcomes data through electronic health records (EHR) even though the treatment protocol will be completed by 96 hours from randomization at the latest. Secondary outcome data will also be collected either during in-person (clinic) visit or via telephone at the 60 and 90-day follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adults of 18 years or older
* Patients hospitalized with a diagnosis of COVID-19 based on central laboratory-confirmed COVID-19 Novel Coronavirus Disease-2019, based on a positive SARS-CoV-2 RT-PCR confirmed within 72 hours prior to enrollment of nasal, oropharyngeal, or BAL specimen with hypoxemia, (i.e., decrease in oxygenation, as outlined below)
* Pulse oximetry saturation (SpO2) < 93% on room air in WHO COVID-19 ordinal scale 3 patients, regardless the need for assisted ventilation, or oxygenation.
* Any new requirement of supplemental oxygen, with any oxygen device (WHO COVID-19 ordinal scale 4-7, regardless of pulse oximetry reading)
* In patients with supplemental oxygen at home, any increase in the requirement of supplemental oxygen.
* In ICU level care

Exclusion Criteria:

* Age less than 18 years
* Known allergy to Vitamin C
* Inability to obtain consent from patient or next of kin
* Presence of diabetic ketoacidosis
* ANY history of oxalate stones at any time
* Patients with Kidney Disease Improving Global Outcomes (KDIGO), CKD stage 4 (eGFR < 30 ml/min, CKD stage 5 and end-stage renal disease on dialysis patients are excluded.
* Patients with Acute Kidney Injury, stage 3.
* Pregnant, or lactating
* Known diagnosis of glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Patients who received the following medications within 7 days prior to enrollment, or plan to receive during enrollment, or 7 days after enrollment: aluminum hydroxide, bortezomib, copper, deferoxamine, amphetamines including derivatives such as fluphenazine.
* Patients with active sickle cell crisis
* Prisoners
* Patients outside ICU level care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alpha (Berry) A Fowler, III, MD, Principal Investigator — Virginia Commonwealth University; Brian Davis, MD, Study Director — Hunter Holmes McGuire VA Medical Center - Richmond, VA
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
There is no default plan to share individual participant data. May be considered upon reaching the VCU IRB

REFERENCES:
- [Background] Dong E, Du H, Gardner L. An interactive web-based dashboard to track COVID-19 in real time. Lancet Infect Dis. 2020 May;20(5):533-534. doi: 10.1016/S1473-3099(20)30120-1. Epub 2020 Feb 19. No abstract available. PMID 32087114
- [Background] Fowler AA 3rd, Truwit JD, Hite RD, Morris PE, DeWilde C, Priday A, Fisher B, Thacker LR 2nd, Natarajan R, Brophy DF, Sculthorpe R, Nanchal R, Syed A, Sturgill J, Martin GS, Sevransky J, Kashiouris M, Hamman S, Egan KF, Hastings A, Spencer W, Tench S, Mehkri O, Bindas J, Duggal A, Graf J, Zellner S, Yanny L, McPolin C, Hollrith T, Kramer D, Ojielo C, Damm T, Cassity E, Wieliczko A, Halquist M. Effect of Vitamin C Infusion on Organ Failure and Biomarkers of Inflammation and Vascular Injury in Patients With Sepsis and Severe Acute Respiratory Failure: The CITRIS-ALI Randomized Clinical Trial. JAMA. 2019 Oct 1;322(13):1261-1270. doi: 10.1001/jama.2019.11825. PMID 31573637
- [Background] Fowler AA 3rd, Fisher BJ, Kashiouris MG. Vitamin C for Sepsis and Acute Respiratory Failure-Reply. JAMA. 2020 Feb 25;323(8):792-793. doi: 10.1001/jama.2019.21987. No abstract available. PMID 32096845
- [Background] Kashiouris MG, L'Heureux M, Cable CA, Fisher BJ, Leichtle SW, Fowler AA. The Emerging Role of Vitamin C as a Treatment for Sepsis. Nutrients. 2020 Jan 22;12(2):292. doi: 10.3390/nu12020292. PMID 31978969
- [Background] Fowler AA 3rd, Syed AA, Knowlson S, Sculthorpe R, Farthing D, DeWilde C, Farthing CA, Larus TL, Martin E, Brophy DF, Gupta S; Medical Respiratory Intensive Care Unit Nursing; Fisher BJ, Natarajan R. Phase I safety trial of intravenous ascorbic acid in patients with severe sepsis. J Transl Med. 2014 Jan 31;12:32. doi: 10.1186/1479-5876-12-32. PMID 24484547
- [Background] Fisher BJ, Seropian IM, Kraskauskas D, Thakkar JN, Voelkel NF, Fowler AA 3rd, Natarajan R. Ascorbic acid attenuates lipopolysaccharide-induced acute lung injury. Crit Care Med. 2011 Jun;39(6):1454-60. doi: 10.1097/CCM.0b013e3182120cb8. PMID 21358394
- [Background] Fisher BJ, Kraskauskas D, Martin EJ, Farkas D, Wegelin JA, Brophy D, Ward KR, Voelkel NF, Fowler AA 3rd, Natarajan R. Mechanisms of attenuation of abdominal sepsis induced acute lung injury by ascorbic acid. Am J Physiol Lung Cell Mol Physiol. 2012 Jul 1;303(1):L20-32. doi: 10.1152/ajplung.00300.2011. Epub 2012 Apr 20. PMID 22523283
- [Background] Fisher BJ, Kraskauskas D, Martin EJ, Farkas D, Puri P, Massey HD, Idowu MO, Brophy DF, Voelkel NF, Fowler AA 3rd, Natarajan R. Attenuation of sepsis-induced organ injury in mice by vitamin C. JPEN J Parenter Enteral Nutr. 2014 Sep;38(7):825-39. doi: 10.1177/0148607113497760. Epub 2013 Aug 5. PMID 23917525
- [Background] Agathocleous M, Meacham CE, Burgess RJ, Piskounova E, Zhao Z, Crane GM, Cowin BL, Bruner E, Murphy MM, Chen W, Spangrude GJ, Hu Z, DeBerardinis RJ, Morrison SJ. Ascorbate regulates haematopoietic stem cell function and leukaemogenesis. Nature. 2017 Sep 28;549(7673):476-481. doi: 10.1038/nature23876. Epub 2017 Aug 21. PMID 28825709
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Infusion | Placebo
Started | 22 | 25
Completed | 22 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infusion | Placebo | Total
Number analyzed (Participants) | 22 | 25 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (13.4) | 60.8 (16.6) | 60.7 (15.0)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  female | 12 | 8 | 20
  male | 10 | 14 | 24
  unknown | 0 | 3 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 21 | 24 | 45
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 8 | 19
  White | 10 | 15 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Weight at Admission (kg) [Mean (Standard Deviation); unit: Kilograms] | 106 (29.5) | 95.3 (30.2) | 100 (30.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in COVID Disease Status
Description: COVID disease status was measured for improvement using the World Health Organization (WHO) ordinal scale for clinical improvement of COVID-19 over ICU admission within 27 days. The WHO scale is a 9-point ordinal scale ranging from uninfected (0), ambulatory (1-2), hospitalized with severe disease (5), hospitalized with intubation and organ support (6-7) and death (score of 8).
Time Frame: Over 27 days from baseline, day 60 and day 90 day
Population: All data points were not available for all subjects at follow-up, Day 27, 60, 90, due to participants not actively being admitted within the ICU and available for assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Infusion | Placebo
Number analyzed (Participants) | 22 | 25
score on a scale
  Baseline (day 0) | 5.09 (0.811) | 5.48 (0.714)
  Day 27: number analyzed (Participants) | 21 | 23
  Day 27 | 3.05 (0.218) | 3.00 (0)
  Day 60: number analyzed (Participants) | 16 | 17
  Day 60 | 3.00 (0) | 2.88 (0.600)
  Day 90: number analyzed (Participants) | 16 | 16
  Day 90 | 3.00 (0) | 2.81 (0.544)

2. Secondary Outcome: Renal Safety Biomarkers - Serum Oxalate
Description: Change in serum oxalate levels
Time Frame: On days 5,7 and 14
Population: Due to staffing/operational challenges in conjunction with only following participants during the ICU admission not all subjects participated in day 5, 7, & 14 oxalate collection. During COVID, methods to limit access to potential exposure & limited PPE restricted collection timepoints. Also, an internal facility error in collection process was noted by outside lab during processing samples. Facility process updated to include new methods, however multiple samples were unable to be processed.
Measure: Mean (Standard Deviation); unit: umol per liter
Arm/Group | Infusion | Placebo
Number analyzed (Participants) | 12 | 21
umol per liter
  Day 5: number analyzed (Participants) | 12 | 18
  Day 5 | 8.96 (9.41) | 10.5 (13.0)
  Day 7: number analyzed (Participants) | 0 | 2
  Day 7 |  | 13.4 (9.48)
  Day 14: number analyzed (Participants) | 0 | 1
  Day 14 |  | 19.0 (0)

3. Secondary Outcome: Renal Safety Biomarkers - Urine Oxalate Stones
Description: Microscopic analysis of urine for presence of oxalate stones
Time Frame: On days 5,7 and 14
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Infusion | Placebo
Number analyzed (Participants) | 12 | 22
Participants
  Day 5: number analyzed (Participants) | 10 | 17
  Day 5 | 1 | 0
  Day 7: number analyzed (Participants) | 1 | 2
  Day 7 | 0 | 0
  Day 14: number analyzed (Participants) | 1 | 3
  Day 14 | 0 | 0

4. Secondary Outcome: Renal Safety Biomarkers - 24-hour Urine Oxalate Levels
Description: Renal safety will be Measured via renal safety biomarkers - 24- hour urine oxalate level
Time Frame: On days 5,7 and 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: umol/day
Arm/Group | Infusion | Placebo
Number analyzed (Participants) | 6 | 7
umol/day
  Day 5: number analyzed (Participants) | 5 | 2
  Day 5 | 40.8 (27.0) | 21.5 (16.3)
  Day 7: number analyzed (Participants) | 0 | 2
  Day 7 |  | 25.5 (6.36)
  Day 14: number analyzed (Participants) | 1 | 3
  Day 14 | 92 | 32.7 (26.7)

5. Secondary Outcome: Acute Kidney Injury-free Days
Description: Renal-failure free days, with AKI defined by the KDIGO criteria
Time Frame: Over 27 days from baseline
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Infusion | Placebo
Number analyzed (Participants) | 22 | 25
Days | 7.36 (8.17) | 8.04 (8.18)

6. Secondary Outcome: Number of Deaths
Description: Mortality by all cause was comprehensively collected using hospital encounter information over 27 days from baseline, in addition to public record review at day 60 and day 90. Results for this outcome represents the number of deaths that have occurred between each time point.
Time Frame: Over 27 days from baseline, day 60 and day 90 day
Measure: Count of Participants; unit: Participants
Arm/Group | Infusion | Placebo
Number analyzed (Participants) | 22 | 25
Participants
  Baseline to Day 27 | 5 | 7
  Day 28 to Day 60 | 0 | 0
  Day 61 to Day 90 | 0 | 0

7. Secondary Outcome: Change in Plasma Ferritin Levels
Description: Difference in plasma ferritin levels in ng/mL, compared to baseline levels
Time Frame: Day 0 (baseline), day 1, day 7
Population: The data is not available for all subjects for all days as reflected in the numbers analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Infusion | Placebo
Number analyzed (Participants) | 22 | 25
ng/mL
  Day 0: number analyzed (Participants) | 22 | 22
  Day 0 | 917 (1350) | 1510 (1500)
  Day 1: number analyzed (Participants) | 19 | 23
  Day 1 | 694 (845) | 1100 (997)
  Day 7: number analyzed (Participants) | 2 | 3
  Day 7 | 638 (488) | 1320 (733)

8. Secondary Outcome: Change in Plasma D-dimer Levels
Description: Difference in D-dimer levels in mcg/mL, compared to baseline levels
Time Frame: Day 0 (baseline), days 1, 2, 3, 4, 5, 6, and 7
Population: Data was not available for all of the subjects for all of the days and therefore was not analyzed as reflected in the numbers.
Measure: Mean (Standard Deviation); unit: mg/L FEU
Arm/Group | Infusion | Placebo
Number analyzed (Participants) | 22 | 25
mg/L FEU
  Baseline: number analyzed (Participants) | 22 | 24
  Baseline | 2.85 (3.45) | 5.60 (6.55)
  Day 1: number analyzed (Participants) | 19 | 22
  Day 1 | 2.65 (2.24) | 5.52 (5.87)
  Day 2: number analyzed (Participants) | 20 | 23
  Day 2 | 2.60 (2.42) | 6.32 (7.04)
  Day 3: number analyzed (Participants) | 16 | 22
  Day 3 | 2.29 (2.18) | 4.99 (5.34)
  Day 4: number analyzed (Participants) | 15 | 21
  Day 4 | 2.71 (2.57) | 3.44 (3.47)
  Day 5: number analyzed (Participants) | 16 | 21
  Day 5 | 2.84 (2.84) | 3.56 (3.49)
  Day 6: number analyzed (Participants) | 12 | 19
  Day 6 | 2.84 (373) | 4.56 (5.18)
  Day 7: number analyzed (Participants) | 5 | 5
  Day 7 | 5.12 (5.26) | 3.80 (4.54)

9. Secondary Outcome: Change in Serum Lactate Dehydrogenase (LDH) Levels
Description: Difference in lactate dehydrogenase (LDH) levels in units/L, compared to baseline levels
Time Frame: Day 0 (baseline), days 1, 2, 3, 4, 5, 6 and 7
Population: Not all of the data was available for all of the subjects as listed below for analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Infusion | Placebo
Number analyzed (Participants) | 22 | 25
mmol/L
  Baseline: number analyzed (Participants) | 22 | 22
  Baseline | 475 (222) | 667 (192)
  Day 1: number analyzed (Participants) | 19 | 22
  Day 1 | 421 (160) | 639 (190)
  Day 2: number analyzed (Participants) | 19 | 23
  Day 2 | 445 (174) | 644 (227)
  Day 3: number analyzed (Participants) | 16 | 21
  Day 3 | 428 (105) | 606 (227)
  Day 4: number analyzed (Participants) | 16 | 22
  Day 4 | 461 (123) | 573 (211)
  Day 5: number analyzed (Participants) | 16 | 21
  Day 5 | 519 (388) | 536 (142)
  Day 6: number analyzed (Participants) | 14 | 19
  Day 6 | 456 (230) | 502 (155)
  Day 7: number analyzed (Participants) | 2 | 3
  Day 7 | 410 (56.6) | 511 (166)

10. Secondary Outcome: Change in Plasma IL-6 Levels
Description: Difference in plasma IL-6 levels in pg/mL, compared to baseline levels
Time Frame: Day 0 (baseline), days 1, 2, 3, 4, 5, 6 and 7
Population: Not all data available for all subjects as indicated below for analysis.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Infusion | Placebo
Number analyzed (Participants) | 22 | 25
pg/mL
  Baseline: number analyzed (Participants) | 22 | 22
  Baseline | 475 (222) | 667 (192)
  Day 1: number analyzed (Participants) | 19 | 22
  Day 1 | 421 (160) | 639 (190)
  Day 2: number analyzed (Participants) | 19 | 23
  Day 2 | 445 (174) | 644 (227)
  Day 3: number analyzed (Participants) | 16 | 21
  Day 3 | 428 (105) | 606 (227)
  Day 4: number analyzed (Participants) | 16 | 22
  Day 4 | 461 (123) | 573 (211)
  Day 5: number analyzed (Participants) | 16 | 21
  Day 5 | 519 (388) | 536 (142)
  Day 6: number analyzed (Participants) | 14 | 17
  Day 6 | 456 (230) | 502 (155)
  Day 7: number analyzed (Participants) | 2 | 3
  Day 7 | 410 (56.6) | 511 (166)

11. Secondary Outcome: Number of Patients Alive and Free of Respiratory Failure
Description: Respiratory failure defined as resource utilization requiring at least 1 of the following: Endotracheal intubation and mechanical ventilation, Oxygen delivered by high-flow nasal cannula (heated, humidified, oxygen delivered via reinforced nasal cannula at flow rates >20L/min with fraction of delivered oxygen ≥0.5), noninvasive positive pressure ventilation, extracorporeal membrane oxygenation
Time Frame: At 28-days
Population: The analyzed population did not reflect all participants still in the study at this time point due to only collecting data for participants remaining in the ICU.
Measure: Count of Participants; unit: Participants
Arm/Group | Infusion | Placebo
Number analyzed (Participants) | 2 | 0
Participants | 2 | 0

12. Secondary Outcome: Number of Patients Alive and Free of Invasive Mechanical Ventilation
Description: Number of patients alive and not requiring invasive mechanical ventilation. The results represent the number of patients who were ventilator free.
Time Frame: At 28-days
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Infusion | Placebo
Number analyzed (Participants) | 2 | 0
Participants | 2 |

ADVERSE EVENTS:
Time Frame: Adverse events were monitored/assessed from baseline to the end of study procedures, or until participants withdrew from the study, up to day 90 for each enrolled participant
Arm/Group | Infusion | Placebo
All-Cause Mortality (participants affected / at risk) | 5/22 | 7/25
Serious Adverse Events (participants affected / at risk) | 0/22 | 1/25
Other Adverse Events (participants affected / at risk) | 0/22 | 3/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infusion (N=22) | Placebo (N=25)
While on study, a subject experienced arrythmia possible ventricular tachycardia (VT) and cardiac ar (Cardiac disorders) | 0 (0) | 1 (1) — While on study, a subject experienced arrythmia possible ventricular tachycardia (VT) and cardiac arrest that resulted in death of the subject on 11NOV2021
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infusion (N=22) | Placebo (N=25)
Vtach episode during study drug infusion (Cardiac disorders) | 0 (0) | 2 (2) — Patient experienced Vtach episode during study drug infusion. Infusion paused, ekg done, study infusion restarted by bedside attending.
Infiltrated IV (General disorders) | 0 (0) | 1 (1) — Swelling at the IV site, removed and reinserted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-10): https://cdn.clinicaltrials.gov/large-docs/84/NCT04344184/Prot_SAP_002.pdf